CLINICAL TRIAL: NCT01149434
Title: Drug- Drug Interaction Study of JI-101 & Everolimus in Advanced Solid Tumors, Expansion Pharmacodynamic Study of JI-101 in Advanced Low Grade Endocrine Tumors, Ovarian Cancers or K-RAS Mutant Colon Cancers
Brief Title: Study of JI-101 in Patients With Advanced Low Grade Endocrine Tumors, Ovarian Cancers or K-RAS Mutant Colon Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of drug efficacy
Sponsor: University of Utah (Other)
Collaborators: Jubilant Innovation Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI43102
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Cancer; Neuroendocrine; Ovarian Cancer; Colon Cancer
Keywords: Low grade endocrine tumors; ovarian cancers; K-RAS mutant colon cancers
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Colonic Neoplasms | interventions — 1-(1-(2-amino-pyridin-4-ylmethyl)-1H-indol-4-yl)-3-(5-bromo-2-methoxyphenyl)urea; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacokinetic Arm (Experimental): Patients going on Pharmacokinetic arm will receive JI-101 & Everolimus (4 patients only)
  Interventions: Drug: JI-101; Drug: Everolimus
- Pharmacodynamic arm (Experimental): Patients going on the Pharmacodynamic study will receive JI-101 only.
  Interventions: Drug: JI-101

INTERVENTIONS:
Drug: JI-101 — JI-101 inhibits angiogenesis, and subsequently tumor growth, by inhibiting three receptor tyrosine kinases: VEGF Receptor Type 2 (VEGFR 2), platelet derived growth factor receptor beta (PDGFR β and Ephrin B4 (EphB4). JI-101 selectively inhibits kinases critical for all three stages of tumor angiogenesis.
Drug: Everolimus — Everolimus is a signal transduction inhibitor that selectively inhibits mTOR (mammalian target of rapamycin), a key and highly conserved serine-threonine kinase, that is present in all cells and is a central regulator of protein synthesis and ultimately cell growth, cell proliferation, angiogenesis, and cell survival. mTOR is the only currently known target of everolimus (1).
  Other Names: RAD001
  Arms: Pharmacokinetic Arm

SUMMARY:
The study consists of two parts: Drug Interaction (Pharmacokinetic) Phase and Pharmacodynamic Phase

The primary study objective for the Drug Interaction Study is to determine the pharmacokinetic interactions between RAD001 and JI-101.

The primary study objective for the Pharmacodynamic Study is progression-free survival at 2 moths, evaluated separately in each of the three cohorts.

These will include a determination of tumor response using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria and an assessment of ephrinB4 expression in blood samples.

Secondary objectives are to determine safety and tolerability of JI-101. The investigational products are everolimus (42-O-(2-hydroxyethyl) rapamycin) and JI-101 (1-[1-(2-amino-pyridin-4-ylmethyl)-1H-indol-4-yl]-3-(5-bromo-2 methoxy-phenyl)-urea)

Eligible patients meeting all study entry criteria will be enrolled in the study. For the Drug Interaction study, patients with solid tumors will receive a single dose (10 mg) of Everolimus by mouth on Day 1 and Day 8 and JI-101 capsules (200 mg) by mouth on Day 8 and Day 15. For the Pharmacodynamic Study, all patients will receive JI-101 capsules by mouth (200 mg BID) for 28 day treatment cycles.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, open-label study to evaluate the safety and efficacy of RAD001 and JI-101 in patients with solid tumors.

Patients will complete all Screening evaluations within 21 days of Study Cycle 1Day 1. All patients will provide written Informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization before any procedures or assessments are initiated for the purposes of the protocol.

For the Drug Interaction Study, Everolimus will be administered to eligible patients at Cycle 1 Day 1 and blood will be drawn for pharmacokinetic analyses prior to dosing and at 0.5, 1, 2, 4, 6, 8, 10, and 24 hours after dosing. On Day 8, Everolimus and JI-101 will be administered and blood will be drawn for pharmacokinetic analyses prior to dosing and at 0.5, 1, 2, 4, 6, 8, 10, and 24 hours after dosing. On Day 15, JI-101 will be administered and blood will be drawn for pharmacokinetic analyses prior to dosing and at 0.5, 1, 2, 4, 6, 8, 10, and 24 hours after dosing. Patients will continue to receive JI-101(200 mg BID) for 28 day treatment cycles. Patients in the Drug Interaction Study will also receive CT scans prior to screening and every 2 treatment cycles.

For the Pharmacodynamic Study, JI-101 will be dispensed to eligible patients at Cycle 1 Day 1. JI-101 will be administered (200 mg BID) for 28 day treatment cycles. PET and CT scans will be performed prior to commencing treatment if it is standard of care. A CT scan will be performed otherwise. Patients will return to the study site every 2 cycles to complete safety assessments with radiologic tumor assessments (CT and/or PET). Adverse events will be monitored following the first administration of investigational product for the duration of the patient's participation in this study. Archival tissue will be collected for detection of mutations in relevant pathways and development of assays to study modulation of pathways that are targeted by JI-101.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age
2. For the Pharmacokinetic Drug Interaction Study: Histologically or cytologically confirmed advanced solid tumors that are refractory to all standard of care therapy or for whom no standard therapy is available, or for whom other standard therapies the patient has denied. For the Pharmacodynamic Study: Histologically or cytologically confirmed metastatic/advanced ovarian carcinoma or metastatic/advanced KRAS mutant colorectal cancer or metastatic/advanced Head and neck squamous cell cancer (HNSCC) that are refractory to all standard therapies therapy or for whom no standard therapy is available, or for whom other standard therapies the patient has denied.
3. At least one measurable tumor as defined by RECIST
4. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
5. Eastern Cooperative Oncology Group (ECOG) of 0 to 2
6. Organ &marrow function as defined in the protocol.
7. No evidence of preexisting uncontrolled hypertension as documented by two baseline blood pressure readings taken at least 1 hour apart
8. Clinically euthyroid
9. Normal range cardiac function
10. For female patients of child-bearing potential, a negative serum pregnancy test at Screening.
11. Current use of an acceptable form of double-barrier birth control
12. Have provided written informed consent

Exclusion Criteria:

1. Known brain or other central nervous system metastases metastases that are not stable for 3 months or longer
2. Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation.
3. Major surgery, radiotherapy, chemotherapy, or cytokine therapy within 28 days of Study Day 0;
4. History of intratumoral bleeding or evidence of bleeding diathesis or coagulopathy
5. Female patients who are pregnant, planning a pregnancy, or who are breastfeeding
6. Known allergy or hypersensitivity to JI-101 or everolimus or any component of the investigational products
7. Use of an investigational drug/device/biologic within 28 days of Study Day 0
8. Current drug or alcohol abuse or history of drug or alcohol abuse within the past two years
9. Known history of or serologic positivity for the Hepatitis B Virus (HBV), or the Hepatitis C Virus (HCV), or for the human immunodeficiency virus (HIV)
10. History of cardiac abnormalities
11. Gastrointestinal (GI) abnormalities
12. Use of concomitant medications that prolong the QT/QTc interval within 14 days prior to Study Day 0
13. History of cerebrovascular accident including transient ischemic attack within the past 6 months
14. History of pulmonary embolism or deep vein thrombosis within the past 6 months
15. History of significant retinopathy or any progressive eye disease that could lead to severe loss of visual acuity or visual field loss during the study period
16. Treatment with heparin or heparin analogs
17. Inability or unwillingness to meet the requirements of the study
18. Other current active malignancy or history of malignancy within the past five years, except for cervical carcinoma in situ, basal cell carcinoma that has been surgically removed, or prostate cancer that is being managed with watchful waiting.
19. Any clinically significant abnormal finding at screening that the investigator judges would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacokinetic Arm Phase 1: Patients going on Pharmacokinetic arm will receive JI-101 & Everolimus (4 patients only)
  JI-101: JI-101 inhibits angiogenesis, and subsequently tumor growth, by inhibiting three receptor tyrosine kinases: VEGF Receptor Type 2 (VEGFR 2), platelet derived growth factor receptor beta (PDGFR β and Ephrin B4 (EphB4). JI-101 selectively inhibits kinases critical for all three stages of tumor angiogenesis.
  Everolimus: Everolimus is a signal transduction inhibitor that selectively inhibits mTOR (mammalian target of rapamycin), a key and highly conserved serine-threonine kinase, that is present in all cells and is a central regulator of protein synthesis and ultimately cell growth, cell proliferation, angiogenesis, and cell survival. mTOR is the only currently known target of everolimus (1).
- Pharmacodynamic Arm Phase 2: Patients going on the Pharmacodynamic study will receive JI-101 only.
  JI-101: JI-101 inhibits angiogenesis, and subsequently tumor growth, by inhibiting three receptor tyrosine kinases: VEGF Receptor Type 2 (VEGFR 2), platelet derived growth factor receptor beta (PDGFR β and Ephrin B4 (EphB4). JI-101 selectively inhibits kinases critical for all three stages of tumor angiogenesis.
Period: Overall Study
Arm/Group | Pharmacokinetic Arm Phase 1 | Pharmacodynamic Arm Phase 2
Started | 4 | 15
Completed | 4 | 10
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Pharmacokinetic Arm - Phase 1: Patients going on Pharmacokinetic arm will receive JI-101 & Everolimus (4 patients only)
  JI-101: JI-101 inhibits angiogenesis, and subsequently tumor growth, by inhibiting three receptor tyrosine kinases: VEGF Receptor Type 2 (VEGFR 2), platelet derived growth factor receptor beta (PDGFR β and Ephrin B4 (EphB4). JI-101 selectively inhibits kinases critical for all three stages of tumor angiogenesis.
  Everolimus: Everolimus is a signal transduction inhibitor that selectively inhibits mTOR (mammalian target of rapamycin), a key and highly conserved serine-threonine kinase, that is present in all cells and is a central regulator of protein synthesis and ultimately cell growth, cell proliferation, angiogenesis, and cell survival. mTOR is the only currently known target of everolimus.
- Pharmacokinetic Arm-Phase II: Patients going on the Pharmacodynamic study will receive JI-101 only.
  JI-101: JI-101 inhibits angiogenesis, and subsequently tumor growth, by inhibiting three receptor tyrosine kinases: VEGF Receptor Type 2 (VEGFR 2), platelet derived growth factor receptor beta (PDGFR β and Ephrin B4 (EphB4). JI-101 selectively inhibits kinases critical for all three stages of tumor angiogenesis.
- Total: Total of all reporting groups
Arm/Group | Pharmacokinetic Arm - Phase 1 | Pharmacokinetic Arm-Phase II | Total
Number analyzed (Participants) | 4 | 15 | 19
Age, Continuous [Mean (Full Range); unit: years] | 72 [65 to 80] | 60 [35 to 79] | 60 [35 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 12
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Effect of JI 101 on Pharmacokinetics Area Under Curve (AUC) (0-inf) of RAD001
Description: Determine the mean percent change that JI-101 has on the peak concentration as determined by calculating the AUC (0-inf) of RAD001 in the presence and absence of JI-101
Time Frame: pre-dose and at 0.5, 1, 2, 4, 6, 8, 10, and 24 hours after dosing (Cycle 1 Day 1 for RAD001 alone and Cycle 1 Day 8 for RAD001 + JI-101
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Pharmacokinetic Arm
Number analyzed (Participants) | 4
percentage change | 165.6 [108.6 to 298.0]

2. Primary Outcome: Effect of RAD001 on Pharmacokinetics AUC(0-inf) of JI-101
Description: Determine the mean percent change that RAD001 has on the peak concentration as determined by calculating the AUC (0-inf) of JI101 in the presence and absence of RAD001
Time Frame: pre-dose and at 0.5, 1, 2, 4, 6, 8, 10, and 24 hours after dosing (Cycle 1 Day 8 for RAD001 + JI101 and Cycle 1 Day 15 for JI-101 alone
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Pharmacokinetic Arm Phase 1
Number analyzed (Participants) | 4
percentage change | 95.3 [89.5 to 137.5]

3. Secondary Outcome: Safety and Tolerability of JI-101
Description: Number of patients experiencing a grade 2 or higher Adverse Event related to JI101
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Pharmacokinetic Arm Phase 1
Number analyzed (Participants) | 4
participants | 4

4. Secondary Outcome: Tumor Response
Description: Response Rate determined by the sum of patients achieving complete or partial response to JI-101 as defined by Response Evaluation Criteria in Solid Tumors. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Pharmacokinetic Arm Phase 1
Number analyzed (Participants) | 4
participants | 0

5. Primary Outcome: Progression Free-Survival in the Ovarian Cancer Cohort
Description: progression-free survival at 2 months. We define progression as using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), to detect a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 months
Population: The intent of this trial was to analyze three different cohorts of patients with different diagnosis. This analysis was conducted with 8 of the enrolled patients that had ovarian disease. Patients enrolled on the remaining cohorts were excluded in this analysis. Results were calculated using Kaplan-Meier product limit methods.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pharmacodynamic Arm Phase 2
Number analyzed (Participants) | 8
percentage of participants | 71.4 [45 to 99]

6. Primary Outcome: Tumor Response in the Ovarian Cancer Cohort
Description: Response Rate determined by the sum of patients achieving complete or partial response to JI-101 as defined by Response Evaluation Criteria in Solid Tumors
Time Frame: 2 years
Population: The intent of this trial was to analyze three different cohorts of patients with different diagnosis. This analysis was conducted with 8 of the enrolled patients that had ovarian disease. The number of patients enrolled on the remaining cohorts were not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Pharmacodynamic Arm Phase 2
Number analyzed (Participants) | 8
Participants | 0

7. Secondary Outcome: Safety and Tolerability of JI-101
Description: Number of patients experiencing a grade 2 or higher Adverse Event related to JI101
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Pharmacodynamic Arm Phase 2
Number analyzed (Participants) | 15
Participants | 12

ADVERSE EVENTS:
Arm/Group | Pharmacokinetic Arm | Pharmacodynamic Arm
Serious Adverse Events (participants affected / at risk) | 1/4 | 4/15
Other Adverse Events (participants affected / at risk) | 4/4 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacokinetic Arm (N=4) | Pharmacodynamic Arm (N=15)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 3 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacokinetic Arm (N=4) | Pharmacodynamic Arm (N=15)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
anemia (Vascular disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 3 (3)
consitpation (Gastrointestinal disorders) | 0 (0) | 1 (1)
dehydration (Gastrointestinal disorders) | 0 (0) | 1 (2)
depression (Nervous system disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (4)
deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Elevated AST (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
fatigue (Investigations) | 2 (2) | 4 (4)
headache (Nervous system disorders) | 0 (0) | 1 (1)
Elevated Alk Phos (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 10 (12)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
left toe infection (Infections and infestations) | 0 (0) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Mouth Soreness (Investigations) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
right upper quadrant pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
weight loss (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No